CLINICAL TRIAL: NCT01602263
Title: Transcranial Direct Current Stimulation (tDCS)and Cognitive Processing
Brief Title: Transcranial Direct Current Stimulation (tDCS) and Cognitive Processing
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00015657; 15657 (Other: Other)
Record Dates: First submitted 2012-05-14; First posted 2012-05-18 (Estimated); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Aphasia; Autism; Schizophrenia
Keywords: Normal cognitive function; Aphasia; Autism; Schizophrenia
MeSH Terms: conditions — Aphasia; Autistic Disorder; Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Controls: Healthy Controls with no known cognitive impairment will have Transcranial Direct Current Stimulation (tDCS) administered and receive either Anodal, Cathodal or Sham tDCS.
  Interventions: Procedure: Transcranial Direct Current Stimulation (tDCS)
- Individuals with schizophrenia: Individuals with schizophrenia and first-degree relatives will have Transcranial Direct Current Stimulation (tDCS) administered and receive either Anodal, Cathodal or Sham tDCS.
  Interventions: Procedure: Transcranial Direct Current Stimulation (tDCS)
- Individuals with aphasia: Individuals with aphasia will have Transcranial Direct Current Stimulation (tDCS) administered and receive either Anodal, Cathodal or Sham tDCS.
  Interventions: Procedure: Transcranial Direct Current Stimulation (tDCS)
- Individuals with high-functioning autism: Individuals with high-functioning autism will have Transcranial Direct Current Stimulation (tDCS) administered and receive either Anodal, Cathodal or Sham tDCS.
  Interventions: Procedure: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Procedure: Transcranial Direct Current Stimulation (tDCS) — Anodal, Cathodal or Sham tDCS.

SUMMARY:
This research is being done to determine whether transcranial direct current stimulation (tDCS) can improve certain mental abilities. In this research, battery powered device is used to deliver very weak electrical current to the surface of the scalp while participants complete cognitive tasks. Our aim is to find out whether tDCS will improve task performance in both healthy adults and those with neurological impairment.

DETAILED DESCRIPTION:
Participants enrolled into this study may be asked to do the following:

* Grant permission for the researchers to view medical records associated with their language/cognitive difficulties (if applicable.
* Complete a questionnaire, provide a health history, and take some pencil-and-paper tests of problem-solving and memory in order to verify eligibility to participate and to able to safely undergo the experimental procedures.
* Complete several tasks (i.e., saying words out loud, naming objects, drawing designs, remembering lists of words, searching for images or letters, and/or completing puzzles) based upon a number of cognitive functions such as language, memory, vision, processing, and perception.
* Wear electrodes that will be placed on the scalp with a large rubberized band. These electrodes will administer very weak electrical current (tDCS) from a battery powered device for 20 to 60 minutes.
* Participation in several study conditions. The exact conditions and their order will be randomized. Under some conditions, participants may receive active stimulation (tDCS) and under other conditions, they may receive sham stimulation.
* The experimental sessions will last approximately 2 hours and participants may be asked to have more than one testing session in a day or to return for additional sessions.
* Have a Magnetic Resonance Imaging (MRI) brain scan.

ELIGIBILITY:
Eligibility Criteria by Study Group

Normal Controls Inclusion Criteria:

* Right handed (as determined by the Edinburgh battery)
* English as native language

Normal Controls Exclusion Criteria:

* Appreciable deficits in hearing
* Appreciable problems with articulation
* Schizophrenia, bipolar disorder, or major depression
* Appreciable accent
* Any neurological disorder associated with cognitive impairment or neuroanatomic abnormality
* Language-based learning disorder
* Any implanted metal device (precludes use of tDCS)
* Any implanted cardiac pacemaker
* Dementia or Mini-Mental State Exam < 24
* Estimated verbal intelligence < 70

Aphasia Group Inclusion Criteria:

* Right handed (as determined by the Edinburgh battery)
* English as native language
* History of acquired left-hemisphere dysfunction

Aphasia Group Exclusion Criteria:

* Appreciable deficits in hearing
* Schizophrenia, bipolar disorder, or major depression
* Appreciable accent
* Language-based learning disorder
* Any implanted metal device
* Any implanted cardiac pacemaker
* Mini-Mental State Exam < 21/27 (omitting naming & items)
* Estimated verbal intelligence < 70

Schizophrenia/First-degree Family Members Inclusion Criteria:

* Right handed (as determined by the Edinburgh battery)
* English as native language
* Diagnosis of schizophrenia (SZ) or bipolar disorder (BD)
* First degree family member of individual with SZ or BD

Schizophrenia/First-degree Family Members Exclusion Criteria:

* Appreciable deficits in hearing
* Appreciable accent
* Any implanted metal device (precludes use of tDCS)
* Any implanted cardiac pacemaker
* Dementia or Mini-Mental State Exam < 24
* Estimated verbal intelligence < 70

High-functioning Autism Inclusion Criteria:

* Right handed (as determined by the Edinburgh battery)
* English as native language
* Diagnosis of High-functioning autism (i.e., Asperger's)

High-functioning Autism Exclusion Criteria:

* Appreciable deficits in hearing
* Schizophrenia, bipolar disorder, or major depression
* Appreciable accent
* Any implanted metal device
* Any implanted cardiac pacemaker
* Dementia or Mini-Mental State Exam < 24
* Estimated verbal intelligence < 70

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: You must also belong to one of three groups to join this study:
  1. Healthy adults with no known deficits in cognition
  2. Adults with acquired language problems (i.e., stroke, mental illness)
  3. Adults with developmental language delays
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2009-01; Primary Completion 2017-12-23 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Indices of cognitive function | The average time frame is 1 hour

SECONDARY OUTCOMES:
Persistence of cognitive enhancements following tDCS | The average time frame is 1 hour
Initiation, endurance and cessation of skin sensations caused by tDCS | The average time frame is 1 hour
  The initiation, endurance and cessation of skin sensations caused by tDCS will be examined in order to develop a more effective blinding procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Gordon, M.D., Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Department of Neurology; Cognitive Neurology/Neuropsychology, Baltimore, Maryland, United States

REFERENCES:
- [Derived] van Steenburgh JJ, Varvaris M, Schretlen DJ, Vannorsdall TD, Gordon B. Balanced bifrontal transcranial direct current stimulation enhances working memory in adults with high-functioning autism: a sham-controlled crossover study. Mol Autism. 2017 Jul 28;8:40. doi: 10.1186/s13229-017-0152-x. eCollection 2017. PMID 28775825
- [Derived] Vannorsdall TD, van Steenburgh JJ, Schretlen DJ, Jayatillake R, Skolasky RL, Gordon B. Reproducibility of tDCS Results in a Randomized Trial: Failure to Replicate Findings of tDCS-Induced Enhancement of Verbal Fluency. Cogn Behav Neurol. 2016 Mar;29(1):11-7. doi: 10.1097/WNN.0000000000000086. PMID 27008245